CLINICAL TRIAL: NCT07097467
Title: Efficacy of Buteyko vs Diaphragmatic Breathing Technique Among the Adolescents With Mouth Breathing Syndrome
Brief Title: Buteyko vs Diaphragmatic Breathing Technique Among the Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Kashish Sahota (Other)
Responsible Party: Sponsor-Investigator, Dr. Kashish Sahota, Assistant Professor, Khalsa College, Amritsar
Organization: Khalsa College, Amritsar (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KCA/PT/2024/958/21
Record Dates: First submitted 2025-07-25; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mouth Breathing Syndrome
Keywords: Breathing techniques; Buteyko vs diaphragmatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Will receive Buteyko Breathing Technique
  Interventions: Other: Buteyko Breathing Technique
- Group B (Active Comparator): Will receive Diaphragmatic breathing technique
  Interventions: Other: Buteyko Breathing Technique

INTERVENTIONS:
Other: Buteyko Breathing Technique — The buteyko breathing technique is a breath holding technique mostly used in Asthma patients

SUMMARY:
This study is about Mouth breathing adolescents. This study is a comparative study between buteyko and diaphragmatic breathing technique to check that which technique is more suitable for mouth breathing children.

DETAILED DESCRIPTION:
The substitution of mouth breathing for nasal breathing or mixed breathing where nose is supplemented by mouth is characterized as mouth breathing syndrome. Mouth breathing results in many facial, occlusal, postural and functional changes. It also has the adverse effect on the memory of young children. Other than that bad breath, sleeping issues are also the major manifestation of mouth breathing syndrome. The buteyko breathing technique has been known to establish the mouth breathing in asthmatic patients and improve their quality of life. This study is to compare the efficacy of both technique among the adolescents with mouth breathing syndrome.

ELIGIBILITY:
Inclusion Criteria:

Mouth Breathing Adolescents, Consented by parents or legal guardians to participate in the study, Mouth breathing syndrome conformed by physician, Positive glatzel mirror test and water test

Exclusion Criteria:

Chronic Respiratory conditions, Neurological conditions, Orthopaedic conditions, Heart diseases, Children undergone tonsillectomy or adenoidectomy, Auditory or visual impairment Body Mass index above 95th percentile

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-06-14 (Actual)

PRIMARY OUTCOMES:
Glatzel Mirror Test | 4 weeks
  A two way mirror is used in this procedure. It is used to determine whether nasal breathing is established or not
Water test | 4 weeks
  Person has to hold the water in mouth for 3 minutes with water closed. It is also used to confirm the mouth breathing

SECONDARY OUTCOMES:
Quality of life ( Mouth Breathing Quality of Life) | 4 weeks
  Mouth Breathing Quality of Life Questionnaire (MBQol) used to check quality if life in mouth breathing children and adolescents.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiotheraoy department, Khalsa College, Amritsar, Punjab, India

IPD SHARING:
Plan to Share IPD: No
All the information is confidential. As per the participants and legal guardian consent form

REFERENCES:
- [Background] Shturman-Ellstein R, Zeballos RJ, Buckley JM, Souhrada JF. The beneficial effect of nasal breathing on exercise-induced bronchoconstriction. Am Rev Respir Dis. 1978 Jul;118(1):65-73. doi: 10.1164/arrd.1978.118.1.65. PMID 677559
- [Background] AbdElmawla Elsaid RA, Zahran WE, Elsaid Hafez DM. Comparison of the Effects of Buteyko and Diaphragmatic Breathing Technique on Improving Pulmonary Functions and Asthma Control among Patients with Bronchial Asthma. Egyptian Journal of Nursing and Health Sciences. 2023 Sep 1;4(3):58-76.
- [Background] Fargaly AA, Bahgat RS, Shrshor SM. Effect of Buteyko Breathing Technique versus Diaphragmatic Breathing on Clinical Outcomes for Children with Lower Respiratory Tract Infection. Tanta Scientific Nursing Journal. 2023 Mar 1;28(1):109-23.
- [Background] Leal RB, Gomes MC, Granville-Garcia AF, Goes PS, de Menezes VA. Impact of breathing patterns on the quality of life of 9- to 10-year-old schoolchildren. Am J Rhinol Allergy. 2016 Sep;30(5):147-52. doi: 10.2500/ajra.2016.30.4363. PMID 27657891
- See also: Occurence of rhinitis, mouth breathing and orofacial alterations in adolescents with asthma — https://www.scielo.br/j/rcefac/a/Gk4xnh58ptzSSqpc9yh6Hkf/?lang=en
- See also: The impact of mouth breathing on dentofacial development: A concise review — https://doi.org/10.3389/fpubh.2022.929165